CLINICAL TRIAL: NCT00003632
Title: A Phase II Study of Intensive Methotrexate and Cytarabine Followed by High Dose Beam Chemotherapy With Autologous Peripheral Blood Progenitor Cell Transplantation in Patients With Newly Diagnosed Primary Central Nervous System Lymphoma
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Newly Diagnosed Central Nervous System Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-086; MSKCC-98086; NCI-G98-1481
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Filgrastim; Carmustine; Cytarabine; Etoposide; Melphalan; Methotrexate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cytarabine
Drug: etoposide
Drug: melphalan
Drug: methotrexate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating patients with newly diagnosed CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy and treatment-related toxicity of high-dose chemotherapy comprising carmustine, etoposide, cytarabine, and melphalan followed by autologous peripheral blood stem cell transplantation in patients with primary central nervous system lymphoma. II. Determine the safety of this regimen in these patients. III. Determine the efficacy of this regimen, in terms of 2-year disease-free survival, in these patients. IV. Assess neurologic outcome using serial neurologic examinations in patients treated with this regimen.

OUTLINE: Induction therapy: Patients receive methotrexate (MTX) IV over 2 hours once on weeks 1, 3, 5, and 7. Patients who respond to treatment receive a fifth dose of MTX on week 9 followed by cytarabine (ARA-C) IV over 3 hours beginning 3 days after completion of MTX infusion and continuing daily for 2 days. Filgrastim (G-CSF) is administered daily beginning 2 days after completion of ARA-C infusion and continuing until harvest of peripheral blood stem cells (PBSC). Patients receive a second course of ARA-C IV beginning 1 month after completion of the first course of ARA-C and continuing daily for 2 days. G-CSF is then administered daily for about 2 weeks. High-dose chemotherapy/transplantation: Patients with stable or responding disease after induction therapy receive high-dose carmustine IV over 1-2 hours on day -7, etoposide IV over 1 hour every 12 hours and ARA-C IV every 12 hours on days -6 to -3, and melphalan IV on day -2. PBSC are reinfused on day 0. Patients receive G-CSF beginning on day 1 and continuing until blood counts recover. Patients are followed monthly for 3 months, every 3 months for 9 months, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed newly diagnosed primary central nervous system (CNS) lymphoma Patients who have inconclusive biopsy or who are not candidates for biopsy may be eligible provided they have a typical cranial MRI or CT scan (presence of hypo, iso, or hyperdense parenchymal contrast-enhancing mass lesions) to insure that leptomeningeal nonparenchymal lymphomas are not included Must meet at least one of the following criteria: Positive CSF cytology for lymphoma or a monoclonal lymphocyte population as defined by cell surface markers Biopsy of the vitreous or uvea demonstrating lymphoma Isolated CNS relapse of systemic non-Hodgkin's lymphoma allowed

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: At least 8 weeks Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT no greater than 2 times upper limit normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: Ejection fraction at least 50% Pulmonary: DLCO at least 50% Other: HIV-1 negative No other active primary malignancy except basal cell skin cancer or carcinoma in situ of the cervix No prior immunodeficiency (e.g., renal transplantation recipient)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for CNS lymphoma Endocrine therapy: Not specified Radiotherapy: No prior cranial irradiation Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-09; Primary Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E. Abrey, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States